CLINICAL TRIAL: NCT00227409
Title: Long-Term Repeated Lead Chelation Therapy in Non-Diabetic Patients With Chronic Renal Insufficiency and High-Normal Body Lead Burden
Brief Title: Long-Term Lead Chelation Therapy and Progressive Renal Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRPG3029; NSC93-2314-B-182A- 079
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2005-09

CONDITIONS: Urologic Disease
Keywords: Repeated chelation therapy; Progressive renal insufficiency; Body lead burden; Long-term outcome; Glomerular filtration rate
MeSH Terms: conditions — Urologic Diseases | interventions — Pentetic Acid

INTERVENTIONS:
Drug: calcium disodium EDTA (edetate calcium disodium)

SUMMARY:
Previous study showed repeated lead chelation therapy significant reduced progressive renal insufficiency in patients with chronic renal diseases and high-normal body lead burden in a placebo-controlled, randomized, 2-year clinical trial, even factors that influence progression, such as blood pressure, the presence or absence of hyperlipidemia, and urinary protein excretion were well controlled.Since relative small sample size and short duration of follow-up were noted in the previous study, whether repeated lead chelation therapy could long-term retard the progression of renal insufficiency remains unknown. Hence, we conducted a 51-month placebo-controlled clinical trial to assess the long-term effect of repeated chelation in progressive renal insufficiency of patients with high-normal body lead burden.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 through 80 years of age who had chronic renal insufficiency were eligible if they had a serum creatinine concentration between 1.5 mg per deciliter (132.6 μmol per liter) and 3.9 mg per deciliter (344.8 μmol per liter), with a decrease in the glomerular filtration rate of less than 5 ml per minute over a period of at least six months
* Blood pressure less than 140/90 mm Hg
* A cholesterol level below 240 mg per deciliter
* Daily protein intake under 1 g per kilogram of body weight
* No known history of exposure to lead or other heavy metals, and a high-normal body lead burden (between 60 and 600 μg, as measured by EDTA mobilization testing and 72-hour urine collection).

Exclusion Criteria:

* Patients who have renal insufficiency with a potentially reversible cause, such as malignant hypertension, urinary tract infection, hypercalcemia, or drug-induced nephrotoxic effects
* Systemic diseases, such as connective-tissue diseases or diabetes mellitus
* Use of drugs that might alter the course of renal disease, such as nonsteroidal anti-inflammatory agents, steroids, or immunosuppressive drugs
* Rapidly progressive glomerulonephritis or a high level of 24-hour urinary protein excretion (more than 8 g per day)
* Previous marked exposure to lead and other metals(lead poisoning or occupational exposure)
* Drug allergies
* Absence of informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11; Study Completion 2005-10

PRIMARY OUTCOMES:
The primary end point was an increase in serum creatinine to 2 times the base-line value or the need for dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ja-Liang Lin, MD, Principal Investigator — Division of Nephrology, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan, China